CLINICAL TRIAL: NCT07190066
Title: Data Collection Campaigns for Early Development Versions of the MELIORA Digital Tools
Brief Title: MELIORA Data Collection Campaigns
Acronym: DCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: BROSTCANCERFORENINGEN AMAZONA I STOCKHOLMS LAN (Unknown); FUNDACION PARA LA INVESTIGACION DEL HOSPITAL CLINICO DE LA COMUNITAT VALENCIANA, FUNDACION INCLIVA (Unknown); Instituto de Investigacion Sanitaria INCLIVA (Other); LIETUVOS SVEIKATOS MOKSLU UNIVERSITETAS (Unknown); PAGALBOS ONKOLOGINIAMS LIGONIAMS ASOCIACIJA (Unknown); SWPS UNIWERSYTET HUMANISTYCZNOSPOLECZNY (Unknown); EUROPEAN FOOD INFORMATION COUNCIL (Unknown); ETHNIKO KENTRO EREVNAS KAI TECHNOLOGIKIS ANAPTYXIS (Unknown); EXUS SOFTWARE MONOPROSOPI ETAIRIA PERIORISMENIS EVTHINIS (Unknown); RISA SICHERHEITSANALYSEN GMBH (Unknown); BIOASSIST SA (Unknown); EUROPEAN HEALTH MANAGEMENT ASSOCIATION (Unknown); ETICAS DATA SOCIETY (Unknown); Karolinska Institutet (Other); PREDICTBY RESEARCH AND CONSULTING S.L. (Unknown)
Responsible Party: Principal Investigator, Yannis Manios, Professor, Harokopio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DCC101136791
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Prevention
Keywords: Behaviors change; Disease prevention; Health behaviour; Primary prevention; Public and environmental health; Breast cancer; Cancer prevention; Sustainable intervention; Nutrition; Diet; Physical activity; Exercise; Lifestyle; Public health; Cancer risk factors; Health communication; Digital health; Health technologies; Artificial intelligence; randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study aims to recruit a total of 300 participants from the four study participating countries to interact with and evaluate the preliminary version of the MELIORA digital app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCC participants (Experimental): Participants will recieve a preliminary version of the MELIORA VCI app
  Interventions: Other: Data Collection campaign

INTERVENTIONS:
Other: Data Collection campaign — Participants will be asked to download the MELIROA app, compatible with iOS and Android, to their smartphones and test it for 14 days. The app will prompt the user to set a weekly goal on physical activity and support daily self-monitoring and step count tracking. Τhe app will also offer culturally adapted educational material through mini-courses, motivational and practical tips and an embedded library of materials relevant to physical activity, healthy diet and alcohol consumption. To boost motivation, it will also include reminders and gamification features like badges and points.

SUMMARY:
To support the development of the MELIORA digital app for the MELIORA main intervention, an initial pilot study (Data Collection Campaign, DCC) is being conducted with the three target participant groups: healthy women at increased risk of developing breast cancer (BC), BC patients, and BC survivors across the four intervention countries (Spain, Greece, Lithuania, Sweden). The planned sample size for each group is 156 healthy women at risk (defined as not meeting recommendations for a healthy lifestyle), 58 BC patients, and 86 BC survivors. Each participant is asked to test and evaluate a preliminary version of the MELIORA app over a 14-day period. The DCC takes place in the early stages of the project, as part of the intervention development phase, to inform the technical refinement and preliminary evaluation of the MELIORA digital app.

DETAILED DESCRIPTION:
The Multimodal Engagement and Sustainable Lifestyle Interventions Optimizing Breast Cancer Risk Reduction Supported by Artificial Intelligence (MELIORA) project addresses the urgent need for innovative, multifaceted approaches to breast cancer (BC) prevention. It promotes sustainable behaviour change through an AI-driven digital intervention. Central to the project is the development and evaluation of the MELIORA Virtual Coach (VC) app, designed to enhance awareness and motivation, and to support healthier lifestyle choices related to physical activity, diet, and alcohol consumption, while also addressing potential implementation barriers.

The overall aim of the Data Collection Campaign (DCC) study is to gather comprehensive socio-demographic, health, lifestyle, and technology-usability data from the project's target participant groups to inform the development and refinement of the MELIORA digital tool and AI algorithms (i.e., the MELIORA app). The specific objectives of the study are to:

* assess the usability of the early version of the MELIORA app and obtain suggestions for further refinement;
* gather user feedback on the relevance, appropriateness, and usefulness of the app's educational content and format;
* inform the design and development of acceptable strategies for behaviour change (e.g., reward strategies);
* further develop AI algorithms for the MELIORA Virtual Coach based on user-provided information.

This DCC pilot study is employing a prospective, exploratory design and is being conducted across four European countries (Greece, Sweden, Spain, and Lithuania) over a 5-month period (from first participant in to last participant out). Recruitment is being carried out through project sites as follows: (i) healthy women at risk of BC in Greece, Spain, and Lithuania; (ii) BC patients in Lithuania and Spain; and (iii) BC survivors in Lithuania and Sweden. The study aims to recruit a total of 300 participants, with target sample sizes of 156 healthy women at risk of BC (defined as not meeting healthy lifestyle recommendations), 58 BC patients, and 86 BC survivors. Participants will test and evaluate a preliminary version of the MELIORA app for 14 days.

Findings from this pilot will provide valuable insights to guide the development of the MELIORA digital tools and AI algorithms, ultimately contributing to improved BC prevention and management through personalised recommendations and interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals residing in Greece, Lithuania, Spain or Sweden.
* Female adults (i.e. ≥18 years of age).
* Ability to understand and complete the outcome measures in one of the participating countries' local languages.
* Ability to provide fully informed consent.
* Having access to and being able to use a smartphone that supports the project app (i.e., iOS or Android smartphone)
* Meeting the criteria for allocation to one of the three following groups:

  * Healthy women with a calculated Βody Μass Ιndex (BMI) ≥ 25 or not meeting the World Health Organization's recommendations of ≥150 minutes of moderate-to-vigorous physical activity per week.
  * Women currently undergoing active treatment for breast cancer or awaiting to begin active treatment for breast cancer.

    * Women survivors of BC having completed active treatment at least six months prior to study enrolment

Exclusion Criteria:

* Inability to provide fully informed consent.
* Inability to understand and communicate in one of the recruitment countries' local languages.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Usability | 14 days
  Assessment of the usability of the first versions of the MELIORA app and users' feedback for further refinement. Participants' experiences and evaluations of the MELIORA app will be collected through a 29-item questionnaire developed for the purposes of the study. Initial questionnaire items were based on the mHealth App Usability Questionnaire (MAUQ) and the Trust in Technology framework, with additional items included to allow evaluations of specific app features. The questionnaire comprises 27 close-ended (with a 1-5 rating Likert scale) and 2 open-ended questions aiming to explore the usability and usefulness of the app, and participants' overall satisfaction with it.
Relevance, appropriateness and usefulness | 14 days
  Users' feedback on the relevance, appropriateness and usefulness of the MELIORA app's educational content and format. Participants will be asked to evaluate the educational materials received, through a pop-up form which will occur at the end of their interaction with each material. The form will contain four questions (with a 1 to 5 rating Likert scale) aiming to gain participants' feedback on the usefulness, relevance, and comprehensibility of the provided materials

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Manios, Professor, Principal Investigator — Department of Nutrition and Dietetics, School of Health Science & Education, Harokopio University, Athens, Greece
Locations (7):
- Harokopio University, Athens, Greece
- Lithuania (2):
  - Lietuvos Sveikatos Mokslų Universitetas (Lsmu), Kaunas
  - Pagalbos Onkologiniams Ligoniams Asociacija (Pola L T), Kaunas
- Spain (2):
  - Fundación Para El Fomento de La Investigación Sanitaria Y Biomédica de La Comunitat Valenciana (Fisabio), Valencia
  - INCLIVA - Instituto de Investigación Sanitaria, Valencia
- Sweden (2):
  - Bröstcancerföreningen Amazona I Stockholms Län (Amazona), Stockholm
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: No
This is a pilot study aiming to gather user feedback to improve the MELIORA digital app to be ready for the main MELIORA intervention.

REFERENCES:
- See also: MELIORA website link — https://melioraproject.eu/